CLINICAL TRIAL: NCT01310218
Title: Length of Postoperative Dressing After Mini-open Carpal Tunnel Release: A Randomized Prospective Comparison
Brief Title: Length of Post Operative Dressing After Carpal Tunnel Release
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UConn Health (Other)
Responsible Party: Craig Rodner MD, Unniversity of Connecticut Health Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCHC 09-158-1; 185190 (Other: UCHC)
Record Dates: First submitted 2011-02-23; First posted 2011-03-08 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-03

CONDITIONS: Carpal Tunnel Syndrome
Keywords: orthopedics, carpal tunnel syndrome, postoperative care
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- extended postoperative dressing (Other): Bulky dressing for 2 weeks
  Interventions: Other: extended postoperative dressing
- short postoperative dressing (Other): 2 day bulky dressing followed by bandaid.
  Interventions: Other: short postoperative dressing

INTERVENTIONS:
Other: extended postoperative dressing — 2 weeks of bulky dressing
  Arms: extended postoperative dressing
Other: short postoperative dressing — 2 days bulky dressing followed by bandaid
  Arms: short postoperative dressing

SUMMARY:
The purpose of the study is to prospectively compare the functional, satisfaction, and wound outcomes of patients treated with one of two accepted methods of postoperative dressing following carpal tunnel release. Hypothesis: There will be no difference between the short term (approximately 2 - 3 days)and longer term (9 to 14 days)bulky dressing groups in terms of outcomes.

ELIGIBILITY:
Inclusion Criteria:

* adults
* carpal tunnel syndrome

Exclusion Criteria:

* previous surgery for Carpal Tunnel Syndrome
* ipsilateral hand, arm, shoulder surgery with continued symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2009-05; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Levine-Katz Scale assessed at different time points. | Levine-Katz Scale at baseline (pre-operation)
  Symptom and function of Carpal Tunnel Syndrome
Change in the Levine-Katz Scale from baseline(pre-operation) at 2 weeks | Baseline and two weeks.
  Symptom and Function of Carpal Tunnel Syndrome
Change in the Levine-Katz Scale from baseline(pre-operation) at 3 months | Baseline and three months.
  Symptom and function of Carpal Tunnel Syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Craig Rodner, MD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States